CLINICAL TRIAL: NCT04442347
Title: A Phase 1b Randomized, Double Blinded, Placebo Controlled, Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of Single Doses of ARCT-810 in Clinically Stable Patients With Ornithine Transcarbamylase Deficiency
Brief Title: Phase 1b Study to Assess Safety, Tolerability, and Pharmacokinetics of ARCT-810 in Stable Adult Subjects With Ornithine Transcarbamylase Deficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arcturus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARCT-810-02
Record Dates: First submitted 2020-06-19; First posted 2020-06-22 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Ornithine Transcarbamylase Deficiency
MeSH Terms: conditions — Ornithine Carbamoyltransferase Deficiency Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blinded, Placebo Controlled
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARCT-810 (Experimental): Ascending single doses of ARCT-810 administered intravenously
  Interventions: Biological: ARCT-810
- Placebo (Placebo Comparator): Single doses of 0.9% Saline administered intravenously
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ARCT-810 — ARCT-810 is an investigational medicinal product comprising Ornithine Transcarbamylase (OTC) mRNA formulated in a lipid nanoparticle (LNP) under development.
  Arms: ARCT-810
Other: Placebo — The placebo for this study is 0.9% sterile saline.
  Arms: Placebo

SUMMARY:
Determine the safety, tolerability and pharmacokinetics of single doses of ARCT-810 in clinically stable patients (stable on standard of care treatment, e.g. diet ± ammonia scavengers) with ornithine transcarbamylase deficiency (OTCD).

DETAILED DESCRIPTION:
This is a single ascending dose study of ARCT-810 in which approximately 12 (up to a maximum of 20) clinically stable patients with ornithine transcarbamylase deficiency (OTCD) are planned to be enrolled.

Each study subject's participation length is approximately 8 weeks, from screening through last study visit. The study comprises an up to 4-week screening period, and a 4-week diet run-in period, to occur concurrently, followed by a 1-day dosing period and a 28-day post-treatment period.

Study participants will be allocated to one of the three single-dose treatment groups (also referred to as cohorts), to test different doses of ARCT-810. Four subjects will be enrolled in each group. Within each cohort, subjects will be randomized 3:1 to receive ARCT-810 or placebo as an IV infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Adequate cognitive ability to consent and recall symptoms over a 1-week time period
2. Males and females ≥18 years of age with documented diagnosis of ornithine transcarbamylase deficiency (OTCD) confirmed with genetic testing, or willing to consent to OTC gene sequencing and deletion/duplication testing
3. Subject's ornithine transcarbamylase deficiency (OTCD) is stable as evidenced by

   1. no clinical symptoms of hyperammonemia AND
   2. an ammonia level <100 µmol/L (170 µg/dL) at the screening evaluation

   Subjects must remain free from symptoms of hyperammonemia throughout the screening period.
4. If using nitrogen ammonia scavenger therapy, must be on a stable regimen (no change in dose or frequency) for ≥ 28 days prior to providing informed consent and throughout the screening period
5. Must have maintained a stable protein-restricted diet (+/- amino acid supplementation) for at least 28 days prior to providing informed consent and continue to maintain a stable diet for the duration of the study
6. Good general health other than OTCD, in the opinion of the Investigator
7. Willing to refrain from strenuous exercise/activity and alcohol for 72 hours before study visits
8. Willingness to comply with procedures and visits
9. Willingness to follow contraception guidelines

Exclusion Criteria:

1. History of clinically significant disease(s), in the opinion of the Investigator
2. Clinically significant screening laboratory values
3. Uncontrolled diabetes
4. Clinically significant anemia
5. Subjects who develop infection during screening must be asymptomatic for at least 7 days prior to dosing
6. Unwillingness to comply with study requirements
7. History of positive HIV, hepatitis C, or chronic hepatitis B
8. Uncontrolled hypertension
9. Malignancy within 5 years prior to study
10. Treatment with another investigational drug, biological agent, or device within 30 days of screening, or 5 half-lives of investigational drug
11. Treatment with any oligonucleotide or mRNA within 6 months of screening, with exceptions for some vaccinations and investigational treatments
12. History of gene therapy, hepatocyte or mesenchymal stem cell transplantation
13. Prior organ transplant
14. History of severe allergic reaction to a liposomal product
15. Recent history of, or current, drug or alcohol abuse
16. Dependence on inhaled (smoked or vaped) or oral cannabis products
17. Systemic corticosteroids within 6 weeks prior to screening
18. Blood donation of 50 to 499 mL within 30 days of screening or of .499 mL within 60 days of screening
19. Other conditions, in the opinion of the Investigator, that would make the subject unsuitable for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence, severity and dose-relationship of adverse events (AEs) | 4 weeks
  Safety and tolerability of ARCT-810 assessed by determining the incidence, severity and dose-relationship of AEs by dose

SECONDARY OUTCOMES:
Change in area under the curve after single dose of ARCT-810 | Up to 4 weeks
  Area under the plasma concentration versus time curve (AUC) from time zero to the last quantifiable time point
Maximum observed plasma concentration (Cmax) after single dose of ARCT-810 | Up to 4 weeks
  The maximum observed plasma concentration (Cmax)
Time at which Cmax occurred after single dose of ARCT-810 | Up to 4 weeks
  The time at which Cmax occurred (Tmax)
AUC0-inf after single dose of ARCT-810 | Up to 4 weeks
  AUC from time zero extrapolated to infinity
AUCExtrap after single dose of ARCT-810 | Up to 4 weeks
  The relative portion of AUC0-inf extrapolated beyond AUC0-t
T1/2 after single dose of ARCT-810 | Up to 4 weeks
  Terminal half-life
MRT0-inf after single dose of ARCT-810 | Up to 4 weeks
  The mean residence time extrapolated to infinity
CL after single dose of ARCT-810 | Up to 4 weeks
  Total body clearance, calculated as dose divided by AUC0-inf
Vss after single dose of ARCT-810 | Up to 4 weeks
  Volume of distribution

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of Florida, Gainesville, Florida
  - M Health Fairview Masonic Children's Hospital, Minneapolis, Minnesota
  - The Mount Sinai Hospital, New York, New York
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Baylor University, Waco, Texas
  - University of Utah, Salt Lake City, Utah
  - Children's Wisconsin - Milwaukee Hospital, Milwaukee, Wisconsin